#### CLINICAL STUDY PROTOCOL

Study Title: An Open-Label, Single-Arm, Historically Controlled, Prospective, Multicenter Phase III Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Immune Globulin Intravenous (Human) GC5107 in Subjects with Primary Humoral Immunodeficiency

SPONSOR: Green Cross Corporation

107 (Mogam Building), Ihyeon-ro 30beon-gil, Giheung-gu, Yongin-si,

Gyeonggi-do, Korea

PROTOCOL NUMBER: GC5107B P3

VERSION 1.0: JANUARY 19, 2016
Date of Amendment 1 February 19, 2016
Date of Amendment 2 March 11, 2016
Date of Amendment 3 March 24, 2016

VERSION 2.0: JUNE 29, 2016
Date of Amendment 1: March 16, 2017
Date of Amendment 2: September 29, 2017
Date of Amendment 3: January 04, 2019

#### **Confidentiality Statement:**

The information contained in this protocol is provided to you in confidence, for review by you, your staff and any applicable regulatory authority or Institutional Review Board/Independent Ethics Committee/Research Ethics Board. It is understood that this information may not be disclosed to any other party in any form without prior authorization from the Sponsor, except to the extent necessary to obtain informed consent from the subject to whom the drug may be administered.

## **SYNOPSIS**

| STUDY TITLE | An Open-Label, Single-Arm, Historically Controlled, Prospective, Multicenter Phase III Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Immune Globulin Intravenous (Human) GC5107 in Subjects with Primary Humoral Immunodeficiency |
|---|---|
| SPONSOR | Green Cross Corporation<br>107 (Mogam BLDG), Ihyeon-ro<br>30beon-gil, Giheung-gu, Yongin-si,<br>Gyeonggi-do, Korea |
| INVESTIGATIONAL<br>PRODUCT | Immune globulin intravenous (human) solution, 10% liquid, GC5107 |
| CLINICAL TRIAL DESIGN | Phase III, open label, single-arm, historically controlled prospective, multicenter study |
| INDICATION AND<br>CLINICAL USE | Treatment of subjects with primary humoral immunodeficiency (PHID) |
| OBJECTIVES | To assess the safety, efficacy, and pharmacokinetics (PK) of GC5107 in subjects with PHID |
| INFUSION RATE | First infusion: Initial rate: 1.0 mg/kg/min (0.01 mL/kg/min) for 30 minutes Incremental rate: • 2.0 mg/kg/min (0.02 mL/kg/min) at 30 minutes • 4.0 mg/kg/min (0.04 mL/kg/min) at 60 minutes • 8.0 mg/kg/min (0.08 mL/kg/min) at 90 minutes If the first infusion is well tolerated, infusions 2-13(17): Initial rate: 2.0 mg/kg/min (0.02 mL/kg/min) for 15 minutes Incremental rate: • 4.0 mg/kg/min (0.04 mL/kg/min) at 15 minutes • 8.0 mg/kg/min (0.08 mL/kg/min) at 30 minutes Maximum rate: 8.0 mg/kg/min (0.08 mL/kg/min) |

| STUDY POPULATION | Male or female aged 2 to 70 years with PHID requiring immune globulin intravenous (IGIV) treatment |
|---|---|
| | • <u>Total Number of Subjects</u> : Up to 50 subjects will be enrolled to obtain at least 42 subjects to be included into the study: |
| | <ul> <li>Adults: at least 26 subjects</li> <li>Adolescents: at least 8 subjects aged ≥ 12 to &lt; 17 years</li> <li>Children: at least 8 subjects aged ≥ 2 to &lt; 12 years</li> </ul> |
| | PK population: at least 20 adult and adolescent subjects |
| | Subjects already stabilized (trough level of 500 mg/dL) on regular IGIV treatment |
| DOSAGE REGIMEN | All subjects will receive intravenous infusions of the investigational product at the same dose and interval as used for their previous IGIV maintenance therapy |
| | Dose of 300 – 900 mg/kg (of body weight) every 21 or 28 days (± 4 days) for 12 months |
| TARGET TROUGH LEVEL | $\geq$ 500 mg/dL (5 g/L) |
| STUDY PERIOD | Approximately 14 months / each subject: |
| | Screening: up to 28 days |
| | • Treatment (investigational product infusions) period: 12 months |
| | • Follow-up period: 3 or 4 weeks |
| INCLUSION CRITERIA | 1. Subject has a confirmed clinical diagnosis of a PHID disease as defined by International Union of Immunological Societies (IUIS) and requires treatment with IGIV, and has documented agammaglobulinemia or hypogammaglobulinemia. |
| | 2. Male or female, aged 2 to 70 years. |
| | 3. The subject has received 300-900 mg/kg of IGIV |
| | therapy at 21(±4 days) or 28(±4 days)day intervals for at least 3 infusion prior to this study. |
| | 4. At least 2 documented IgG trough levels of |
| | ≥ 500 mg/dL are obtained at two infusion cycles |

 $(21(\pm 4 \text{ days}) \text{ or } 28(\pm 4 \text{ days}) \text{ days})$  within 12 months prior to study treatment. 5. Subject is willing to comply with all requirements of the protocol. 6. Females of child-bearing potential with a negative pregnancy test at screening and females who agree to employ adequate birth control measures during the study. 7. Males who agree to practice adequate birth control measures during the study. 8. Subject, parent or guardian has signed the informed consent form and an assent form for children ( $\geq 2$  to < 12 years of age at study entry) and adolescents  $( \ge 12 \text{ to} < 17 \text{ years of age at study entry})$  as appropriate per study documentation and regulations of the local jurisdiction. 9. Authorization to access personal health information. 10. Subject currently participating in a clinical trial with another experimental IGIV may be enrolled if he/she has received stable IGIV therapy for at least 3 infusion cycles prior to receiving GC5107 and all inclusion and exclusion criteria are satisfied. Other IGIVs will be prohibited for an infusion cycle (21(±4 days) or 28(±4 days) days) prior to the first infusion of GC5107 until the completion of Follow-up visit. 11. Subject currently participating in a trial of subcutaneous immunoglobulin (SCIG) can be enrolled if he/she is switched to IGIV for three infusion cycles  $(21(\pm 4 \text{ days}) \text{ or } 28(\pm 4 \text{ days}) \text{ days})$  prior to enrollment in this study. 1. Subject has secondary immunodeficiency. **EXCLUSION CRITERIA** 2. Subject was newly diagnosed with PHID and has not yet been treated with immunoglobulin. 3. Subject has been diagnosed with dysgammaglobulinemia or isolated IgG subclass deficiency or isolated IgA deficiency with known anti-IgA antibodies.

**Green Cross Corporation** 

Protocol Number: GC5107B P3

- Green Cross Corporation Protocol Number: GC5107B\_P3
- 4. History of severe reaction or hypersensitivity to IGIV or other injectable forms of IgG.
- 5. Subject has a lifetime history of at least one thrombotic event including deep vein thrombosis, cerebrovascular accident, pulmonary embolism, transient ischemic attacks, or myocardial infarction.
- 6. Subject has received blood products other than human albumin or human immunoglobulin within 12 months prior to enrollment.
- 7. Subject has protein losing enteropathy, nephrotic syndrome or lymphangiectasia.
- 8. Subject has had clinical signs or symptoms of an acute infection within 7 days prior to screening.
- 9. Subject has a known history or is positive at enrollment for HIV type 1/2 by nucleic acid testing (NAT), hepatitis B virus (HBsAg and NAT), hepatitis C virus (by NAT), or hepatitis A virus (by NAT).
- 10. Subject has levels of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times of the upper limit of normal for the laboratory designated for the study.
- 11. Subject has profound anemia (hemoglobin [Hgb]  $\leq 8 \text{ g/dL}$ ) or persistent severe neutropenia ( $\leq 1000 \text{ neutrophils per mm}^3$ ).
- 12. Subject has a severe chronic condition such as renal failure (creatinine concentration > 2.0 times the upper limit of normal), congestive heart failure (New York Heart Association III/IV), cardiomyopathy, cardiac arrhythmia associated with thromboembolic events (e.g., atrial fibrillation), unstable or advanced ischemic heart disease, hyperviscosity, or any other condition that the investigator believes is likely to interfere with evaluation of the investigational product or with satisfactory conduct of the trial.
- 13. Subject has a history of a malignant disease, other than properly treated carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin within 24 months prior to enrollment.
- 14. Subject has history of epilepsy or migraines not completely controlled by medication.

| | 15. Subject is receiving the following medication: |
|---|---|
| | • Corticosteroids (oral or parenteral daily dose of ≥ 0.15 mg/kg/day of prednisone or equivalent). |
| | Other immunosuppressive drugs or chemotherapy. |
| | 16. Females who are pregnant, breast feeding or planning a pregnancy during the study. Women who become pregnant during the study will be withdrawn from the study. Males who do not agree to use contraception will not qualify to be enrolled in the study. Males are not allowed to donate sperm during the study. |
| | 17. Subject has participated in another clinical study within 3 weeks prior to study enrollment. |
| EFFICACY ENDPOINT | 1) Primary Efficacy Endpoint: The incidence of acute serious bacterial infections meeting Food and Drug Administration (FDA) guidance criteria (bacterial pneumonia, bacteremia/sepsis, bacterial meningitis, visceral abscess, osteomyelitis/septic arthritis). |
| | 2) Secondary Efficacy Endpoints |
| | • The incidence of infections other than acute serious bacterial infections meeting FDA guidance criteria. |
| | The number of days missed from work/school/kindergarten/daycare, or days unable to perform normal daily activities due to infections. |
| | • The number of days that the care provider of the pediatric subject had to miss work in order to care for the child due to infections. |
| | The number days of unscheduled physician visits due to infections. |
| | • The number of days of hospitalizations due to infections. |
| | • The number of days of intravenous (IV) therapeutic antibiotics. |
| | The number of days of oral therapeutic antibiotics. |
| | Time to resolution of infections. |
| | • The incidence of infections other than serious bacterial infections by trough IgG levels. |
| SAFETY ENDPOINTS | 1) Primary Safety Endpoint: The proportion of infusions with temporally associated adverse events |

(AEs) that occur during or within 1 hour, 24 hours, and 72 hours following an infusion of investigational product (including AEs that were determined to be unrelated to the product). 2) Secondary Safety Endpoints • The overall incidence of all AEs that occur during or within 1 hour, 24 hours ,and 72 hours following an infusion of investigational product. • The frequency of all AEs that occur during the study regardless of the investigator's assessment of their relationship to investigational product. • The frequency of suspected adverse reactions as defined by all AEs either classified by investigator or sponsor as at least possibly related to GC5107. • Changes in vital signs, physical examinations, and laboratory test results. • The number and proportion of GC5107 infusions for which the infusion rate was decreased due to AEs. • The proportion of AEs considered by the investigator to be investigational product related. safety from Viral (freedom transmission blood-borne viral diseases): human the immunodeficiency virus (HIV) 1&2, hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), and parvovirus B19. **PHARMACOKINETIC** 1) Primary PK Endpoints **ENDPOINTS** • PK parameters of total IgG (assessed in PK population). • Trough serum total IgG levels before each infusion of GC5107 in all subjects and the interval between infusions will be recorded. 2) Secondary PK Endpoints • PK parameters of IgG subclasses (assessed in PK population) • Trough serum level of IgG subclasses and specific IgG antibodies before Infusion 1, 5, 9, 13 (for 28-day infusion subject) or Infusion 1, 5, 11, 17 (for 21-day infusion subject) o anti-Hemophilus influenza type b

**Green Cross Corporation** 

Protocol Number: GC5107B P3

anti-Streptococcus pneumonia serotypes anti-Tetanus toxoid o anti-Cytomegalovirus (CMV) • Number and proportion of subjects who failed to meet the target IgG trough level (500 mg/dL) at any time point equal to or subsequent to 5th infusion (estimated 5 half-lives). ANALYTICAL PLAN / Efficacy data will be evaluated by comparing the number STATISTICAL METHOD of acute serious bacterial infections per subject per year according to the FDA guideline of an upper one-sided 99% confidence limit < 1.0 per subject per year. The primary safety endpoint will be analyzed with the objective of demonstrating that the percentage of infusions with one or more infusion-related ΑE is less than Pharmacokinetic parameters (clearance, mean residence time, volume of distribution, and terminal half-life) will be noncompartmental estimated by fitting individually to the data for each subject in the PK population, except for the AUC which will be determined using a (log-) trapezoidal rule as the area above the previous trough level. Pharmacokinetic parameters will be derived from serum IgG levels and presented descriptively. Trough levels of IgG subclasses will be summarized relative to dosing interval. All other data will be reported descriptively.

**Green Cross Corporation** 

Protocol Number: GC5107B P3

# **Authorization Page**

| Protocol Title | An Open-Label, Single-Arm, Historically Controlled, Prospective, Multicenter Phase III Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Immune Globulin Intravenous (Human) GC5107 in Subjects with Primary Humoral Immunodeficiency |
|---|---|
| Protocol<br>Number | GC5107B_P3 |
| Version | V 2.0 Amendment 3 |
| Sponsor | |

#### **Table of Contents**

| CLINI | CAL STUDY PROTOCOL | 1 |
|--------|-------------------------------------------------------|----|
| SYNOF | PSIS | 2 |
| AUTH | ORIZATION PAGE | 9 |
| TABLE | E OF CONTENTS | 10 |
| LIST O | OF TABLES | 13 |
| LIST O | OF ABBREVIATIONS | 14 |
| 1. | INTRODUCTION | 16 |
| 1.1. | BACKGROUND: PRIMARY HUMORAL IMMUNODEFICIENCY DISEASES | |
| 1.2 | Non-clinical Data | |
| 1.3 | BENEFIT/RISK STATEMENT | |
| 1.4 | RATIONALE | |
| 1.5 | GCP COMPLIANCE | 19 |
| 1.6 | STUDY POPULATION | 19 |
| 2. | STUDY OBJECTIVE | 19 |
| 2.1. | Primary Efficacy Endpoint | |
| 2.2. | SECONDARY EFFICACY ENDPOINTS | 19 |
| 2.3. | Primary Safety Endpoint | 20 |
| 2.4. | SECONDARY SAFETY ENDPOINTS | 20 |
| 2.5. | PRIMARY PHARMACOKINETIC ENDPOINTS | 21 |
| 2.6. | SECONDARY PHARMACOKINETIC ENDPOINTS | 21 |
| 3. | INVESTIGATIONAL PLAN | 21 |
| 3.1. | DURATION OF THE STUDY | |
| 3.2. | INVESTIGATORS AND STUDY CENTERS | 22 |
| 3.3. | RANDOMIZATION AND STRATIFICATION | 22 |
| 3.4. | Blinding | 22 |
| 4. | SELECTION OF STUDY POPULATION | 22 |
| 4.1. | Inclusion Criteria | 23 |
| 4.2. | Exclusion Criteria | 24 |
| 4.3. | WITHDRAWAL OF SUBJECTS | |
| 4.4. | EARLY DISCONTINUATION OF STUDY | |
| 4.5 | STOPPING RULES | 27 |
| 5. | STUDY CONDUCT | 27 |
| 5.1. | Treatment Regimens | 27 |
| 5.2. | Treatment Assignment | 27 |
| 5.3. | SUBJECT IDENTIFICATION | 27 |
| 5.4. | PHYSICAL EXAMINATION | 28 |
| 5.5. | MEDICAL HISTORY AND DEMOGRAPHY | |
| 5.6. | Subject Diary | |
| 5.7. | DOSAGE | |
| 5.8. | VISIT SCHEDULE | |
| 5. | .8.1 Screening: Day -28 or -21 to Day -1 | 30 |

| | <i>5.8.2</i> | First Infusion (Day 1, Week 0) | 31 |
|---|---|---|---|
| | 5.8.3 | Safety Visit (72 hours after the end of first infusion) | 32 |
| | 5.8.4 | Second Infusion (Week 3 of 21-day and Week 4 of 28-day Infusion Schedules) | 33 |
| | 5.8.5 S | afety Visit (72 hours after the end of second infusion) | 34 |
| | 5.8.6 | Third to 17th Infusion (21-day Schedule); 3rd to 13th Infusion (28-day Schedule) | 34 |
| | 5.8.7 | Additional Tests | |
| | 5.8.8 | PK Analysis: 5th Infusion of All Participating Subjects | 36 |
| | 5.8.10 | Follow-up | |
| | 5.8.11 | Unscheduled Visit Procedures | 36 |
| į | 5.9 In | IVESTIGATIONAL PRODUCT PREPARATION AND HANDLING | 37 |
| į | 5.10 In | FUSION RATES | 38 |
| | 5.11 Pr | RODUCT DESCRIPTION | 39 |
| | | ABELING AND PACKAGING | |
| ļ | 5.13 SH | HIPMENT AND STORAGE | 39 |
| | 5.14 Co | DNCOMITANT MEDICATIONS | 40 |
| | 5.14.1 | the state of the s | |
| | | Prohibited Medications | |
| | 5.15 In | VESTIGATIONAL PRODUCT ACCOUNTABILITY AND DOCUMENTATION | 41 |
| | 5.16 Di | ESTRUCTION OF USED AND UNUSED INVESTIGATIONAL PRODUCT | 41 |
| 5. | Δ | SSESSMENT OF EFFICACY | 42 |
| | | RIMARY EFFICACY ENDPOINT: INCIDENCE OF ACUTE SERIOUS BACTERIAL INFECTION | |
| | | CONDARY EFFICACY ENDPOINTS | |
| 7. | | SSESSMENT OF PHARMACOKINETICS | |
| | | G TROUGH LEVELS | |
| | | G SUBCLASSES/SPECIFIC ANTIBODIES – TROUGH LEVELS | |
| | 7.3. Pi | HARMACOKINETIC PARAMETERS OF TOTAL IGG AND SERUM LEVELS OF IGG SUBCLASSES | 45 |
| 3. | A. | SSESSMENT OF SAFETY | 46 |
| 8 | 8.1. SA | IFETY PARAMETERS | 46 |
| | 8.1.1 | Vital Signs | 46 |
| | 8.1.2 | Routine blood tests | 47 |
| | 8.1.3 | Other safety laboratory parameters | 48 |
| 8 | 8.2. Ai | OVERSE EVENTS | 48 |
| | 8.2.1 | Definition of an Adverse Event (AE) | |
| | 8.2.2 | Adverse Reaction | 49 |
| | 8.2.3 | Suspected Adverse Reaction | |
| | 8.2.4 | Unexpected Adverse Events | |
| | 8.2.5 | Serious Adverse Event (SAE) | |
| 8 | | OCUMENTATION OF ADVERSE EVENTS | |
| 8 | 8.4. As | SSESSMENT OF ADVERSE EVENTS | 52 |
| | 8.4.1 | Assessment of Severity | 52 |
| | | ssessment of Causality | |
| | | EPORTING SERIOUS ADVERSE EVENTS | |
| | | RUG SAFETY MONITORING BOARD | |
| 8 | 8.7. W | ARNINGS AND PRECAUTIONS | 56 |
| | 5.7. VV | | |
| 9. | | FATISTICAL METHODS AND SAMPLE SIZE | |
| 9. | S | TATISTICAL METHODS AND SAMPLE SIZE | 57 |
| | <b>S</b> 7<br>9.1. St | ATISTICAL DESIGN/METHOD | . <b> 57</b><br>57 |
| | S | | . <b> 57</b><br>57 |

| 9.1.4 Primary Efficacy Endpoints 55 9.1.5 Secondary Efficacy Endpoints 66 9.1.6 Pharmacokinetic Endpoints 62 9.1.7 Safety Endpoints 62 9.2. Level of Significance 66 9.3. STATISTICAL SOFTWARE 65 10. ETHICS 63 10.1. INVESTIGATIONAL REVIEW BOARD/RESEARCH ETHICS BOARD 65 10.2. INFORMED CONSENT AND ASSENT 65 10.3. CONFIDENTIALITY 66 10.4. DECLARATION OF HELSINKI 65 11. QUALITY CONTROL AND QUALITY ASSURANCE 65 11.1. GENERAL INFORMATION 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 66 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 66 15. LIABILITIES AND INSURANCE 66 16. REFERNCES 69 17. APPENDICES 74 PRINCIPAL INVESTIGATOR'S AGREEMENT 75 | 9.1. | 3 Demographics | 59 |
|---|---|---|---|
| 9.1.6 Pharmacokinetic Endpoints 66 9.1.7 Safety Endpoints 62 9.2. Level of Significance 62 9.3. STATISTICAL SOFTWARE 63 10. ETHICS 63 10.1 Investigational Review Board/Research Ethics Board 63 10.2 Informed Consent and Assent 63 10.3 Confidentiality 64 10.4 Declaration of Helsinki 65 11. QUALITY CONTROL AND QUALITY ASSURANCE 65 11.1. General Information 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 66 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 69 16. REFERNCES 69 17. APPENDICES 74 | 9.1. | | |
| 9.1.7 Safety Endpoints | 9.1. | | |
| 9.2. Level of Significance 62 9.3. STATISTICAL SOFTWARE 63 10. ETHICS 63 10.1. Investicational Review Board/Research Ethics Board 63 10.2. Informed Consent and Assent 63 10.3. Confidentiality 64 10.4. Declaration of Helsinki 65 11. QUALITY CONTROL AND QUALITY ASSURANCE 65 11.1. General Information 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 9.1. | | |
| 9.3. STATISTICAL SOFTWARE 63 10. ETHICS 63 10.1. INVESTIGATIONAL REVIEW BOARD/RESEARCH ETHICS BOARD 65 10.2. INFORMED CONSENT AND ASSENT 65 10.3. CONFIDENTIALITY 64 10.4. DECLARATION OF HELSINKI 65 11. QUALITY CONTROL AND QUALITY ASSURANCE 65 11.1. GENERAL INFORMATION 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | | | |
| 10. ETHICS 63 10.1. INVESTIGATIONAL REVIEW BOARD/RESEARCH ETHICS BOARD 63 10.2. INFORMED CONSENT AND ASSENT 63 10.3. CONFIDENTIALITY 64 10.4. DECLARATION OF HELSINKI 65 11. QUALITY CONTROL AND QUALITY ASSURANCE 65 11.1. GENERAL INFORMATION 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 66 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | | | |
| 10.1. INVESTIGATIONAL REVIEW BOARD/RESEARCH ETHICS BOARD 65 10.2. INFORMED CONSENT AND ASSENT 65 10.3. CONFIDENTIALITY 64 10.4. DECLARATION OF HELSINKI 65 11. QUALITY CONTROL AND QUALITY ASSURANCE 65 11.1. GENERAL INFORMATION 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 9.3. | STATISTICAL SOFTWARE | 63 |
| 10.1. INVESTIGATIONAL REVIEW BOARD/RESEARCH ETHICS BOARD 65 10.2. INFORMED CONSENT AND ASSENT 65 10.3. CONFIDENTIALITY 64 10.4. DECLARATION OF HELSINKI 65 11. QUALITY CONTROL AND QUALITY ASSURANCE 65 11.1. GENERAL INFORMATION 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 10. | ETHICS | 63 |
| 10.3. CONFIDENTIALITY 64 10.4. DECLARATION OF HELSINKI 65 11. QUALITY CONTROL AND QUALITY ASSURANCE 65 11.1. GENERAL INFORMATION 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 10.1. | | |
| 10.4. DECLARATION OF HELSINKI 65 11. QUALITY CONTROL AND QUALITY ASSURANCE 65 11.1. GENERAL INFORMATION 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 10.2. | INFORMED CONSENT AND ASSENT | 63 |
| 11. QUALITY CONTROL AND QUALITY ASSURANCE 65 11.1. GENERAL INFORMATION 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 10.3. | CONFIDENTIALITY | 64 |
| 11.1. GENERAL INFORMATION 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 10.4. | DECLARATION OF HELSINKI | 65 |
| 11.1. GENERAL INFORMATION 65 11.2. QUALITY CONTROL BY THE MONITORING TEAM 65 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM 65 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 11. | OUALITY CONTROL AND OUALITY ASSURANCE | 65 |
| 11.3. QUALITY ASSURANCE BY AN AUDIT TEAM | 11.1. | GENERAL INFORMATION | 65 |
| 12. DATA HANDLING AND RECORD KEEPING 66 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 11.2. | QUALITY CONTROL BY THE MONITORING TEAM | 65 |
| 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 11.3. | QUALITY ASSURANCE BY AN AUDIT TEAM | 65 |
| 12.1. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS 66 12.2. DATA COLLECTION AND MANAGEMENT 66 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 12. | DATA HANDLING AND RECORD KEEPING | 66 |
| 12.3. RECORD KEEPING 67 13. CHANGES IN THE CONDUCT OF THE STUDY 67 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 12.1. | | |
| 13. CHANGES IN THE CONDUCT OF THE STUDY | 12.2. | DATA COLLECTION AND MANAGEMENT | 66 |
| 14. REPORTING AND PUBLICATION 68 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 74 | 12.3. | RECORD KEEPING | 67 |
| 15. LIABILITIES AND INSURANCE 68 16. REFERNCES 69 17. APPENDICES 74 | 13. | CHANGES IN THE CONDUCT OF THE STUDY | 67 |
| 16. REFERNCES | 14. | REPORTING AND PUBLICATION | 68 |
| 17. APPENDICES | 15. | LIABILITIES AND INSURANCE | 68 |
| | 16. REF | ERNCES | 69 |
| PRINCIPAL INVESTIGATOR'S AGREEMENT75 | <b>17. APP</b> | ENDICES | 74 |
| | PRINCIF | PAL INVESTIGATOR'S AGREEMENT | 75 |

## **List of Tables**

| Table 1: Study Timeline | 30 |
|---------------------------------------------------------------------|----|
| Table 2: Infusion rates for GC5107 | 38 |
| Table 3: Mean Infection Rates and Power of Study Sample Size | 58 |
| Table 4: Schedule of Subject Evaluations - 28 Day Infusion Schedule | |
| Table 5: Schedule of Subject Evaluations – 21 Day Infusion Schedule | |

# **List of Abbreviations**

| AE | Adverse event |
|-----------|-----------------------------------------------------|
| AIDS | Acquired immune deficiency syndrome |
| ALT | Alanine aminotransferase |
| AMS | Aseptic Meningitis Syndrome |
| AST | Aspartate aminotransferase |
| AUC | Area under the curve |
| BAL | |
| | Bronchoalveolar lavage |
| BP | Blood pressure |
| BUN | Blood urea nitrogen |
| bw | Body weight |
| °C | Degrees Celsius |
| CK | Creatine kinase |
| CL | Total body clearance |
| $C_{max}$ | Maximum concentration |
| $C_{min}$ | Minimum concentration |
| CMV | Cytomegalovirus |
| CPMP | Committee for Proprietary Medicinal Products |
| CR | Clinical Research |
| CRF | Case report form |
| CRO | Contract Research Organization |
| CSF | Cerebrospinal fluid |
| CT | Computed tomography |
| CVID | Common variable immunodeficiency |
| D5W | Dextrose 5 % in water |
| DAT | Direct Antiglobulin (Coombs) test |
| DSMB | Drug Safety Monitoring Board |
| EU | European Union |
| °F | Degrees Fahrenheit |
| FDA | Food and Drug Administration |
| g | Gram |
| GCP | Good Clinical Practice |
| GLP | Good Laboratory Practice |
| GMP | Good Manufacturing Practice |
| h | Hour |
| HAV | Hepatitis A virus |
| HBV | Hepatitis B virus |
| HCV | Hepatitis C virus |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | Human immunodeficiency virus |
| ICF | Informed consent form |
| ICH | International Conference on Harmonization |
| IDF | Immune Deficiency Foundation |
| IDL | minute Deficiency Foundation |

| IgA | Immunoglobulin A |
|---|---|
| IgG | Immunoglobulin G |
| IGIV | Immunoglobulin intravenous |
| IgM | Immunoglobulin M |
| IP | Investigational product |
| IRB | Institutional Review Board |
| ITP | Immune Thrombocytopenic Purpura |
| ITT | Intention-to-treat |
| IV | Intravenous |
| Kg | Kilogram |
| L | Liter |
| LDH | Lactate dehydrogenase |
| MedDRA | Medical dictionary for regulatory activities |
| mg | Milligram |
| min | Minute |
| mL | Milliliter |
| MRI | Magnetic resonance imaging |
| No. | Number |
| NSAID | Non-steroidal anti-inflammatory drugs |
| NYHA | New York Heart Association |
| PCR | Polymerase chain reaction |
| PHID | Primary humoral immunodeficiency |
| PI | Principal investigator |
| PK | Pharmacokinetic |
| PO | Oral |
| PP | Per protocol |
| PPS | Per protocol data set |
| QA | Quality Assurance |
| QC | Quality Control |
| RBC | Red Blood Cells |
| SAE | Serious adverse event |
| SCIG | Subcutaneous immunoglobulin |
| t <sub>1/2</sub> | Elimination half-life |
| t <sub>max</sub> | Time point of maximum concentration (C <sub>max</sub> ) |
| TRALI | Transfusion related acute lung injury |
| USA | United States of America |
| ULN | Upper limit of normal |
| WBC | White blood cell |
| WHO | World Health Organization |
